CLINICAL TRIAL: NCT03710876
Title: A Phase 3, Open-Label, Randomized, Parallel Group Study to Evaluate the Efficacy and Safety of Intrapleural Administration of Adenovirus-Delivered Interferon Alpha-2b (rAd-IFN) in Combination With Celecoxib and Gemcitabine in Patients With Malignant Pleural Mesothelioma
Brief Title: Efficacy & Safety of rAd-IFN Administered With Celecoxib & Gemcitabine in Patients With Malignant Pleural Mesothelioma
Acronym: INFINITE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Ventures Limited (Industry)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rAd-IFN-MM-301; 2017-003169-82 (EudraCT Number)
Record Dates: First submitted 2018-06-22; First posted 2018-10-18 (Actual); Results first posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-04

CONDITIONS: Malignant Pleural Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Gemcitabine; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Active Comparator): rAd-IFN (Study Day 1) + celecoxib (Study Days 1 to 14) + gemcitabine (Study Days 14 and 21 [i.e., Days 1 and 8 of the first gemcitabine treatment cycle], gemcitabine will be administered on a 21-day cycle, unless the cycle is modified due to toxicity/delay, and repeated every 3 weeks until disease progression/early termination [ET]
  Interventions: Biological: rAd-IFN; Drug: Celecoxib Oral Product; Drug: Gemcitabine
- Control Group (Placebo Comparator): Celecoxib (Study Days 1 to 14) + gemcitabine (Study Days 14 and 21 [i.e., Days 1 and 8 of the first gemcitabine treatment cycle], gemcitabine will be administered on a 21-day cycle, unless the cycle is modified due to toxicity/delay, and repeated every 3 weeks until disease progression/ET.
  Interventions: Drug: Celecoxib Oral Product; Drug: Gemcitabine

INTERVENTIONS:
Biological: rAd-IFN — Adenovirus-Delivered Interferon Alpha-2b
  Other Names: Nadofaragene firadenovec
  Arms: Treatment Group
Drug: Celecoxib Oral Product — 400 mg twice daily
  Other Names: COX II Inhibitor
Drug: Gemcitabine — 1250 mg/m2 administered intravenously on Days 1 and 8 of a 21-day cycle and continued every 3 weeks until disease progression/ early termination
  Other Names: Chemotherapy

SUMMARY:
This study will evaluate intrapleural administration of Adenovirus-Delivered Interferon Alpha-2b (rAd-IFN) in combination with Celecoxib and Gemcitabine in patients with histologically confirmed Malignant Pleural Mesothelioma (MPM) who have failed a minimum of 1 treatment regimen and a maximum of 2 treatment regimens, 1 of which must have been an anti-folate and platinum combination regimen.

Eligible patients will be randomized 1:1 to either:

1. Treatment group: rAd-IFN + Celecoxib followed by Gemcitabine
2. Control group: Celecoxib followed by Gemcitabine

Patients randomized to the treatment group will receive rAd-IFN administered into the pleural space via an Intrapleural catheter (IPC) or similar intrapleural device on study Day 1.

The primary objective of this study is to compare the overall survival (OS) associated with rAd IFN, when administered with celecoxib and gemcitabine, versus that associated with celecoxib and gemcitabine alone for the treatment of patients with MPM

DETAILED DESCRIPTION:
TITLE: A Phase 3, Open-Label, Randomized, Parallel Group Study to Evaluate the Efficacy and Safety of Intrapleural Administration of Adenovirus-Delivered Interferon Alpha-2b (rAd-IFN) in Combination with Celecoxib and Gemcitabine in Patients with Malignant Pleural Mesothelioma

PROTOCOL NUMBER: rAd-IFN-MM-301

STUDY DRUGS: Nadofaragene firadenovec (Recombinant adenovirus vector containing the human interferon alpha-2b gene: rAd-IFN), celecoxib, and gemcitabine

PHASE: 3

INDICATION: Malignant pleural mesothelioma (MPM)

SPONSOR: Ferring Ventures Ltd.

SITES: Up to 45 sites globally

OBJECTIVES:

The primary objective of this study is to compare the overall survival (OS) associated with rAd IFN, when administered with celecoxib and gemcitabine, versus that associated with celecoxib and gemcitabine alone for the treatment of patients with MPM who have failed a minimum of 1 treatment regimen and a maximum of 2 treatment regimens, 1 of which must have been an anti-folate and platinum combination regimen.

The secondary objectives of this study are:

* To compare between rAd-IFN, when administered with celecoxib and gemcitabine, versus that associated with celecoxib and gemcitabine alone for the treatment of patients with MPM who have failed a minimum of 1 treatment regimen and a maximum of 2 treatment regimens, 1 of which must have been an anti-folate and platinum combination regimen, with respect to:

  * Survival rate at 12 months and every 6 months thereafter;
  * Progression-free survival (PFS);
  * Best response (complete response, partial response, or stable disease); and
  * Safety of rAd-IFN; and
* To evaluate rAd-IFN, when administered with celecoxib and gemcitabine, in a sub-set of patients with MPM who have failed a minimum of 1 treatment regimen and a maximum of 2 treatment regimens, 1 of which must have been an anti-folate and platinum combination regimen, with respect to viral shedding and biodistribution.

The exploratory objectives of this study are:

• To compare between rAd-IFN, when administered with celecoxib and gemcitabine, versus that associated with celecoxib and gemcitabine alone for the treatment of patients with MPM who have failed a minimum of 1 treatment regimen and a maximum of 2 treatment regimens, 1 of which must have been an anti-folate and platinum combination regimen, with respect to:

* Health-related Quality-of-Life,
* The relationship between immunological status and response to treatment, and
* Biocorrelates of response to treatment.

POPULATION:

The population for this study is patients with histologically confirmed MPM of epithelioid or biphasic (predominantly [>50%] epithelioid) histology who have failed a minimum of 1 treatment regimen and a maximum of 2 treatment regimens, 1 of which must have been an anti-folate and platinum combination regimen.

STUDY DESIGN AND DURATION:

The study is an open-label, randomized, parallel group study conducted in patients with MPM and confirmed epithelioid or biphasic histology (if biphasic, histology must be predominantly [>50%] epithelioid) who have received a minimum of 1 treatment regimen and a maximum of 2 treatment regimens, 1 of which must have been an anti-folate and platinum combination regimen.

Screening assessments must be completed within 28 days prior to Study Day 1, and eligible patients will be randomized to either:

1. Treatment group: rAd-IFN (Study Day 1) + celecoxib (Study Days 1 to 14) + gemcitabine (Study Days 14 and 21 [i.e., Days 1 and 8 of the first gemcitabine treatment cycle], gemcitabine will be administered on a 21-day cycle, unless the cycle is modified due to toxicity/delay, and repeated every 3 weeks until disease progression/early termination [ET]); or
2. Control group: celecoxib (Study Days 1 to 14) + gemcitabine (Study Days 14 and 21[i.e., Days 1 and 8 of the first gemcitabine treatment cycle], gemcitabine will be administered on a 21-day cycle, unless the cycle is modified due to toxicity/delay, and repeated every 3 weeks until disease progression/ET).

Treatment Phase Patients randomized to receive rAd-IFN (treatment group) will have an intrapleural catheter (IPC) or similar device either previously in place or inserted for the study, permitting drug administration to an accessible pleural space. The rAd-IFN will be diluted to a volume of 25 mL using sterile normal saline and will be administered directly to the pleural space via the IPC or similar device.

The IPC or similar device will then be flushed with up to 20 mL of sterile normal saline.

Patients will receive gemcitabine until disease progression/ET. All adverse events will be captured from the time of the main study's informed consent through 30 days after the last dose of study treatment (rAd-IFN, celecoxib, and/or gemcitabine). All treatment emergent adverse events (TEAEs) and serious adverse events (SAEs) will be followed until resolution or stabilization.

Clinical Follow-Up Phase Following disease progression/ET, patients in the rAd-IFN treatment group will be followed every 6 months (±14 days) for survival and safety for up to 5 years after receiving the first dose of rAd-IFN, assuming consent has not been withdrawn. All previously recorded TEAEs and SAEs will be followed until resolution or stabilization. Patients in the control group will not continue in the clinical Follow-up phase and study participation will conclude after end of study treatment.

DOSAGE FORMS AND ROUTE OF ADMINISTRATION:

Patients randomized to the treatment group will receive rAd-IFN (3 × 1011 viral particles) on Study Day 1, diluted to a total volume of 25 mL using sterile normal saline and administered into the pleural space via an IPC or similar device. The IPC or similar device will then be flushed with up to 20 mL of sterile normal saline.

All study patients (treatment and control) will receive:

* Celecoxib administered at a dose of 400 mg twice daily orally on Study Days 1 to 14; and
* Gemcitabine starting on Study Day 14, using the following treatment regimen: 1250 mg/m2 administered intravenously on Days 1 and 8 of a 21-day gemcitabine cycle, unless the cycle is modified due to toxicity/delay, and continued every 3 weeks until disease progression/ET.

STATISTICAL ANALYSES:

The primary analysis of the primary endpoint is a comparison of the OS curves between the 2 treatment groups using a log-rank test. A Cox proportional hazards model with treatment as an explanatory variable will be used to assess the magnitude of the treatment difference in OS. The hazard ratio and the associated 95% confidence interval obtained from the Cox proportional hazards model will be presented.

The median OS and the 95% confidence interval for each treatment group will be estimated using the Kaplan-Meier method and summarized by treatment group. Plots of the Kaplan-Meier curve of OS will be presented by treatment group.

Secondary analyses of the primary endpoint will include a comparison of the survival rates at various time points since randomization.

Secondary time-to-event endpoints will be analysed in the same manner as the primary efficacy endpoint.

Categorical efficacy endpoints will be summarized and compared between groups using Fisher's exact test.

The nature, incidence, severity, relatedness, expectedness, seriousness, and outcome of TEAEs will be summarized by treatment group for safety analyses.

SAMPLE SIZE DETERMINATION:

The planned sample size is approximately 50 patients. The sample size is not based on statistical considerations. Patient recruitment into the study has been significantly slower than expected due to several technical study challenges. Therefore, Trizell has decided to discontinue screening and enrolment into the study after a total of approximately 50 patients have been randomized to treatment. It is anticipated that approximately 44 events (equivalent to 89% of the planned 50 enrolled patients) will be observed 24 months after the last patient is randomized. The final analysis of the study will be conducted after the forty-fourth event (death) or 30 months after the last patient is randomized, whichever occurs first.

DATA AND SAFETY MONITORING BOARD:

An independent Data and Safety Monitoring Board (DSMB) will be convened for this study to monitor safety, efficacy, and study integrity. All aspects of the DSMB's scope of review and procedures will be detailed in a DSMB charter.

ELIGIBILITY:
Inclusion Criteria

Patients who meet all of the following criteria will be eligible to participate in the study:

1. Aged 18 years or older at the time of consent;
2. Able to give informed consent;
3. Has a confirmed histological diagnosis of MPM with histological type epithelioid or biphasic (if biphasic, histology must be predominantly [50%] epithelioid). Histological diagnosis of MPM will be confirmed centrally using specimens or slides from tumor specimens obtained at the time of initial presentation or a subsequent procedure. Central confirmation of diagnosis with immunohistochemistry will be performed, and independent central confirmation will be required for study entry;
4. Measurable disease, per modified Response Evaluation Criteria in Solid Tumors [RECIST] 1.1 (see Section 7) for pleural mesothelioma;
5. Has received a minimum of 1 treatment regimen and a maximum of 2 treatment regimens, which may have been chemotherapeutic and/or immunotherapeutic treatment regimens for MPM which included at least 1 anti-folate and platinum combination regimen;

   * Adjuvant or neoadjuvant therapy represent 1 line of therapy each;
   * Patients who have undergone primary surgical resection and/or radiation therapy to the pulmonary site are eligible to participate. For clarity, surgical resection and/or radiation therapy to the pulmonary site are not exclusionary and are not considered a line of therapy;
   * Treatment that is split between pre-surgical resection and post-surgical resection and is the same regimen will be counted as 1 regimen. Patients meeting this condition should be discussed with the Medical Monitor prior to including the patient in the study;
6. Has a pleural space accessible for IPC or similar device insertion. Patients with a previously inserted IPC or similar device may be enrolled, and the pre-existing IPC or similar device can be used for vector administration as long as it is functional and has no evidence of local infection;
7. Life expectancy 12 weeks in the judgement of the Investigator;
8. Eastern Cooperative Oncology Group (ECOG) status of 1 or 0;
9. Female and male patients:

   * Female patients of childbearing potential must have a negative pregnancy test upon entry into this study and agree to use a highly effective method of contraception from Screening until 1 month after the last dose of gemcitabine;

     * Highly effective methods of contraception that result in a low failure rate (i.e., <1% per year) when used consistently and correctly include combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, or transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, or implantable), intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomized partner, or sexual abstinence;
     * True abstinence, when in line with the preferred and usual lifestyle of the patient, is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of study participation and for 1 month after the last dose of gemcitabine. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, and post-ovulation method) and withdrawal are not acceptable methods of contraception; and
   * Female patients of non-childbearing potential must be either postmenopausal (no menstrual period for a minimum of 12 months) or surgically sterile upon entry into the study;
   * Male patients must be either surgically sterile or agree to use a double-barrier contraception method from Screening until 6 months after the last dose of gemcitabine; o Where available and in accordance with local practice, male patients must be advised to seek further advice regarding cryoconservation of sperm prior to gemcitabine treatment due to the possibility of infertility after therapy with gemcitabine; and
10. Adequate laboratory values at Screening:

    * Hemoglobin 9 g/dL;
    * White blood cell count 3500/µL;
    * Absolute neutrophil count 1500/µL;
    * • Platelet count 100,000/µL;
    * International normalized ratio (INR) and activated partial thromboplastin time (aPTT) below the upper limit of normal (ULN). It is expected that patients receiving anticoagulation therapy will not have INR and aPTT results that fall within normal limits. It is not intended to exclude these patients and, therefore, medical discretion is permitted for patients who have clinically acceptable results in regards to their current concomitant anticoagulant therapy;
    * Aspartate aminotransferase (AST) 3 × ULN;
    * Alanine aminotransferase (ALT) 3 × ULN;
    * Total bilirubin 2 × ULN;
    * Estimated glomerular filtration rate (calculated using the Modification of Diet in Renal Disease study equation [see Appendix B]) 50 mL/min/1.73 m2; and
    * Serum albumin 2.5 g/dL.

Exclusion Criteria

Patients who meet any of the following criteria will be excluded from participation in the study:

1. Is "treatment-naïve" (i.e., has not received at least 1 anti-folate and platinum combination regimen);
2. Has previously received 3 or more lines of systemic chemotherapeutic or immunotherapeutic treatment. Treatment that is split between pre-surgical resection and post-surgical resection and is the same regimen will be counted as 1 regimen. Patients meeting this condition should be discussed with the Medical Monitor prior to including the patient in the study;
3. Has previously received treatment with gemcitabine;
4. Has stage IV extrathoracic metastatic disease;
5. Inadequate pulmonary function of clinical significance as per Investigator review;
6. Clinically significant pericardial effusion (i.e., as judged by the Investigator and/or requiring drainage) detected by computed tomography (CT) scan at Screening. Standard of care CT scans completed within 2 weeks prior to Screening may be used in place of the Screening CT scan on a case by-case basis as agreed with the Medical Monitor;
7. Prior therapy(ies), if applicable, must be completed according to the criteria below prior to vector administration:

   * Cytotoxic chemotherapy, at least 21 days from last dose;
   * Non-cytotoxic chemotherapy (e.g., small molecule inhibitor), at least 14 days from last dose;
   * Monoclonal antibody, at least 30 days from last dose;
   * Non-antibody immunotherapy (e.g., tumor vaccine), at least 42 days from last dose;
   * Radiotherapy, at least 14 days from last local site radiotherapy;
   * Hematopoietic growth factor, at least 14 days from last dose; or
   * Study drug, 30 days or 5 half-lives, whichever is longer, from last dose;
8. Patient previously treated with IFNs (e.g., for chronic active hepatitis);
9. Suspected/known hypersensitivity to IFN-α2b or rAd-IFN (including any of its excipients);
10. Known hypersensitivity to celecoxib (including any of its excipients) or sulfonamides;
11. Known hypersensitivity to gemcitabine (including any of its excipients);
12. Impaired cardiac function or clinically significant cardiac disease including the following:

    * New York Heart Association class III or IV congestive heart failure;
    * Myocardial infarction within the last 12 months; and
    * Patients known to have impaired left ventricular ejection fraction per institutional standards and of clinical significance as per Investigator review;
13. Women who are pregnant or breastfeeding;
14. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, depression, or psychiatric illness/social situations within the last 12 months;
15. Patients with active, known, or suspected auto-immune disease or a syndrome that requires systemic or immunosuppressive agents (oral prednisolone or equivalent at a dose of 10 mg per day is permitted); NOTE: patients with vitiligo, residual hypothyroidism due to auto immune disease only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll;
16. History of asthma, acute rhinitis, nasal polyps, angioneurotic edema, urticaria, or other allergic type reactions after taking acetylsalicylic acid or NSAIDs, including COX-2 inhibitors;
17. History of ulcer disease or gastrointestinal bleeding;
18. Uncontrolled or poorly controlled hypertension (i.e., blood pressure >160/100 mmHg) requiring 3 or more anti-hypertensive drugs;
19. Heart rate corrected QT interval using Fridericia's formula >470 ms on resting 12-lead electrocardiogram (ECG);
20. Patients receiving lithium;
21. Any significant disease which, in the opinion of the Investigator, would place the patient at increased risk of harm if he/she participated in the study;
22. History of a prior malignancy for which treatment was completed <2 years prior to Screening or for which the patient has continued evidence of disease, or concurrent malignancy that is clinically unstable and requires tumor-directed treatment;
23. Has a congenital or acquired immunodeficiency, including patients with known history of infection with human immunodeficiency virus;
24. Has both serum albumin 2.5 to 3.5 g/dL and total bilirubin >1.5 ULN;
25. History of clinically significant inflammatory bowel disease requiring systemic (parenteral) immunosuppressive therapy within 5 years prior to Screening; or
26. History of galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2026-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Sterman, MD, Principal Investigator — NYU Langone Laura and Isaac Perlmutter Cancer Center
Locations (29):
- United States (7):
  - University of California, Los Angeles (UCLA) - Medical Center, Los Angeles, California
  - University of California, San Francisco (UCSF), San Francisco, California
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Marlene & Stewart Greenbaum Comprehensive Cancer Center, Baltimore, Maryland
  - University of Maryland Medical Center, Baltimore, Maryland
  - Masonic Cancer Center - University of Minnesota, Minneapolis, Minnesota
  - University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania
- Australia (2):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Monash Medical Centre, Clayton, Victoria
- Institut Universitaire de Cardiologie et de Pneumologie De Quebec, Québec, Sainte-Foy, Canada
- France (7):
  - Institut Bergonie, Bordeaux
  - CHRU de Brest - Hopital Augustin Morvan, Brest
  - CHU de Caen - Hopital Cote de Nacre, Caen
  - CHRU de Lille, Lille
  - Institut Curie - Oncologie Medicale, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Nantes - Hôpital Nord Laennec, Saint-Herblain
- Germany (2):
  - Evangelisches Krankenhaus Hamm, Hamm
  - Universitatsklinikum Regensburg, Regensburg
- Azienda Ospedaliero Universitaria Senese, Cancer Immunotherapy, Siena, Tuscany, Italy
- Poland (2):
  - Med Polonia Sp. z o.o., Poznan
  - Centrum Onkologii Instytut im. Marii Sklodowskiej - Curie, Klinika Nowotworow Tkanek Miekkich, Kosci i Czerniakow, Warsaw
- Russia (2):
  - Petrov National Medical Research Center of Oncology, Saint Petersburg
  - Volgograd Regional Clinical Oncology Dispensary, Volgograd
- United Kingdom (5):
  - Derriford Hospital ; Derriford Hospital, Plymouth, Devon
  - Beatson, West of Scotland Cancer Centre, Glasgow, Scotland
  - Royal Marsden Foundation Trust, Sutton, Surrey
  - Guy's and St. Thomas' NHS Trust, London
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to recruitment in January 2019 and was scheduled to complete recruitment by May 2021, with a target of approximately 300. 53 patients were randomized to treatment.
Period: Overall Study
Arm/Group | Treatment Group | Control Group
Started | 27 | 26
Treated | 27 | 22
Completed | 27 | 22
Not Completed | 0 | 4
Not completed — Death | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: All patients who were appropriately randomized into the study and who received at least 1 dose of study drug (rAd-IFN, celecoxib, or gemcitabine).
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Control Group | Total
Number analyzed (Participants) | 27 | 26 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 6 | 10
  >=65 years | 23 | 20 | 43
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.5 (8.84) | 69.3 (10.08) | 70.9 (9.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 20 | 22 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 25 | 20 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  Canada | 1 | 1 | 2
  United States | 6 | 7 | 13
  Poland | 2 | 4 | 6
  United Kingdom | 7 | 4 | 11
  Italy | 1 | 0 | 1
  Australia | 1 | 1 | 2
  France | 8 | 7 | 15
  Germany | 1 | 0 | 1
  Russia | 0 | 2 | 2
Overall Number of Baseline Participants [Count of Participants; unit: Participants] | 27 | 26 | 53

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Time to death (from any cause) from randomization
Time Frame: 4 years and 8 months
Population: The Full Analysis Set, which comprised all patients who were appropriately randomized into the study and who received at least 1 dose of study drug (rAd-IFN, celecoxib, or gemcitabine).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 27 | 22
Months | 17.6 [8.3 to 31.8] | 15.5 [9.2 to 16.6]
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Test type: Superiority; p = 0.2840, Log Rank — 1-sided; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.43 to 1.59]

2. Secondary Outcome: Progression Free Survival
Description: Time measured in months, from randomization to the time when the modified Response Evaluation Criteria in Solid Tumour criteria for disease progression are first met, or when death from any cause occurs
Time Frame: 4 years and 8 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 27 | 22
Months | 7.4 [4.1 to 14.2] | 14.6 [4.1 to 15.8]

3. Secondary Outcome: Best Response: Objective Response Rate (ORR)
Description: Best overall response (BOR) was defined as the best response designation, in the order of Complete Response (CR), Partial Response (PR), Stable Disease (SD), Progressive Disease (PD), or Not Evaluable (NE), for each patient that was recorded between the date of randomization and the date of documented disease progression per mRECIST or mRECIST version 1.1, or the date of subsequent anticancer therapy or cancer-related surgery (i.e., surgical resection of tumour), whichever occurred first. ORR was defined as the proportion of patients with a BOR of CR or PR.
Time Frame: 4 years and 8 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 27 | 22
Participants | 2 | 1
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Test type: Superiority; p = 1.0000, Fisher Exact — 2-sided; Risk Difference (RD) = 2.9, 95% CI 2-sided [-17.3 to 24.3] — Risk difference is proportion achieving objective response in r+C+G group minus the proportion achieving objective response in C+ G group. The confidence interval was calculated by the exact conditional method of Chan and Zhang

4. Secondary Outcome: Best Response: Disease Control Rate (DCR)
Description: Disease control rate (DCR) was defined as the proportion of patients with a BOR of CR, PR, or Stable Disease (SD).
Time Frame: 4 years and 8 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 27 | 22
Participants | 19 | 15
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Test type: Superiority; p = 1.0000, Fisher Exact; Risk Difference (RD) = 2.2, 95% CI 2-sided [-25.2 to 29.2] — Risk difference is proportion achieving response in r+C+G group minus the proportion achieving response in C+ G group. The confidence interval was calculated by the exact conditional method of Chan and Zhang

5. Secondary Outcome: Best Response: Clinical Benefit Rate (CBR)
Description: Clinical Benefit Rate (CBR) was defined as the proportion of patients with a BOR of CR, PR, or SD >/= 6 months.
Time Frame: 4 years and 8 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 27 | 22
Participants | 9 | 9
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Test type: Superiority; p = 0.7665, Fisher Exact; Risk Difference (RD) = -7.6, 95% CI 2-sided [-34.9 to 20.3] — [estimate comment as in outcome 4, analysis 1]

6. Other Pre Specified Outcome: Survival Rate at 12 Months
Description: Proportion surviving at 12 months
Time Frame: 12 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of survivors
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 27 | 22
Percentage of survivors | 59.3 [38.6 to 75.0] | 63.6 [40.3 to 79.9]
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Percentage proportion calculated by Kaplan-Meier method; Test type: Superiority; p = 0.7537, Chi-squared — 2-sided; Variance calculated by Greenwood's method; Risk Difference (RD) = -4.4, 95% CI 2-sided [-31.7 to 23.0] — Risk difference is estimated probability of survival in r+C+G minus the estimated probability of survival in C+G group

7. Other Pre Specified Outcome: Survival Rate at 18 Months
Description: Proportion surviving at 18 months
Time Frame: 18 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of survivors
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 27 | 22
Percentage of survivors | 48.1 [28.7 to 65.2] | 29.8 [12.4 to 49.5]
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Percentage proportion calculated by Kaplan-Meier method; Test type: Superiority; p = 0.1855, Chi-squared — 2-sided; Variance calculated by Greenwood's method; Risk Difference (RD) = 18.4, 95% CI 2-sided [-8.8 to 45.6] — Risk difference is estimated probability of survival in r+C+G minus the estimated probability of survival in C+G group

8. Other Pre Specified Outcome: Survival Rate at 24 Months
Description: Proportion surviving at 24 months
Time Frame: 24 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of survivors
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 27 | 22
Percentage of survivors | 37.0 [19.6 to 54.6] | 24.8 [9.2 to 44.3]
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Percentage proportion calculated by Kaplan-Meier method; Test type: Superiority; p = 0.3570, Chi-squared — 2-sided; Variance calculated by Greenwood's method; Risk Difference (RD) = 12.2, 95% CI 2-sided [-13.8 to 38.3] — Risk difference is estimated probability of survival in r+C+G minus the estimated probability of survival in C+G group

9. Other Pre Specified Outcome: Survival Rate at 30 Months
Description: Proportion surviving at 30 months
Time Frame: 30 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of survivors
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 27 | 22
Percentage of survivors | 33.3 [16.8 to 50.9] | 19.8 [6.3 to 38.9]
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Percentage proportion calculated by Kaplan-Meier method; Test type: Superiority; p = 0.2856, Chi-squared — 2-sided; Variance calculated by Greenwood's method; Risk Difference (RD) = 13.5, 95% CI 2-sided [-11.3 to 38.3] — Risk difference is estimated probability of survival in r+C+G minus the estimated probability of survival in C+G group

10. Other Pre Specified Outcome: Survival Rate at 36 Months
Description: Proportion surviving at 36 months
Time Frame: 36 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of survivors
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 27 | 22
Percentage of survivors | 25.9 [11.5 to 43.1] | 19.8 [6.3 to 38.9]
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Percentage proportion calculated by Kaplan-Meier method; Test type: Superiority; p = 0.6173, Chi-squared — 2-sided; Variance calculated by Greenwood's method; Risk Difference (RD) = 6.1, 95% CI 2-sided [-17.8 to 30.0] — Risk difference is estimated probability of survival in r+C+G minus the estimated probability of survival in C+G group

11. Other Pre Specified Outcome: Survival Rate at 42 Months
Description: Proportion surviving at 42 months
Time Frame: 42 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of survivors
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 27 | 22
Percentage of survivors | 25.9 [11.5 to 43.1] | 19.8 [6.3 to 38.9]
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Percentage proportion calculated by Kaplan-Meier method; Test type: Superiority; p = 0.6173, Chi-squared — 2-sided; Variance calculated by Greenwood's method; Risk Difference (RD) = 6.1, 95% CI 2-sided [-17.8 to 30.0] — Risk difference is estimated probability of survival in r+C+G minus the estimated probability of survival in C+G group

12. Other Pre Specified Outcome: Adverse Events Grade 3 or 4.
Description: To evaluate the number of patients with Common Terminology Criteria for Adverse Events Grade 3 or 4.
Time Frame: 4 years and 8 months.
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 27 | 22
Participants | 18 | 17

ADVERSE EVENTS:
Time Frame: The Safety Analysis Set comprises all patients who received at least 1 dose of study drug (rAd-IFN, celecoxib, or gemcitabine), from study start on 27 August 2019 to Data Cut-off on 07 May 2024, a period of 4 years and 8 months.
Description: Standard (S)AE definitions. The Intent-to-Treat (ITT) Analysis Set comprised all randomized patients; this represents the population for the calculation of All-Cause Mortality.
  The Safety Analysis Set comprised all patients who received at least 1 dose of study drug; this represents the population for presentation of the Adverse Events data.
Arm/Group | Treatment Group | Control Group
All-Cause Mortality (participants affected / at risk) | 22/27 | 19/26
Serious Adverse Events (participants affected / at risk) | 10/27 | 12/22
Other Adverse Events (participants affected / at risk) | 27/27 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=27) | Control Group (N=22)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 2 (4)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Pleural infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary opedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 0 (0)
Spinal cord injury thoracic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=27) | Control Group (N=22)
Fatigue (General disorders) | 11 (27) | 8 (20)
Pyrexia (General disorders) | 4 (7) | 6 (12)
Asthenia (General disorders) | 8 (27) | 4 (5)
Oedema peripheral (General disorders) | 6 (8) | 5 (9)
Non-cardiac chest pain (General disorders) | 3 (3) | 1 (1)
Chest pain (General disorders) | 2 (3) | 1 (1)
Malaise (General disorders) | 0 (0) | 2 (2)
Cather site extravasation (General disorders) | 2 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (16) | 8 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 11 (34) | 9 (18)
Neutropenia (Blood and lymphatic system disorders) | 5 (10) | 6 (17)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 2 (4)
Leukopenia (Blood and lymphatic system disorders) | 2 (3) | 1 (3)
Thrombocytosis (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 17 (39) | 7 (12)
Constipation (Gastrointestinal disorders) | 4 (4) | 6 (7)
Vomiting (Gastrointestinal disorders) | 6 (8) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (7) | 1 (1)
Abdominal distention (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dyspep[sia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (5) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 4 (5) | 2 (2)
Neutrophil count decreased (Investigations) | 4 (5) | 4 (10)
White blood cell count decreased (Investigations) | 2 (14) | 4 (9)
Gamma-glutamyltransferase increased (Investigations) | 2 (3) | 3 (5)
Amylase increased (Investigations) | 2 (2) | 2 (2)
Blood creatinine increased (Investigations) | 0 (0) | 4 (4)
Platelet count decreased (Investigations) | 2 (7) | 2 (7)
Weight decreased (Investigations) | 0 (0) | 4 (4)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 3 (10)
Lipase increased (Investigations) | 2 (6) | 1 (2)
Lymphocyte count decreased (Investigations) | 2 (7) | 1 (1)
Body temperature increased (Investigations) | 2 (3) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 6 (9) | 6 (9)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (4) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (3) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (2) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (7)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (2)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (5) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 2 (3) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 2 (3)
Cystitis (Infections and infestations) | 2 (4) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 2 (6) | 2 (2)
Headache (Nervous system disorders) | 4 (5) | 0 (0)
Lethargy (Nervous system disorders) | 2 (2) | 1 (2)
Insomnia (Psychiatric disorders) | 2 (2) | 3 (3)
Depression (Psychiatric disorders) | 1 (1) | 3 (3)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 5 (5) | 0 (0)
Proteinuria (Renal and urinary disorders) | 3 (11) | 2 (9)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 2 (12) | 3 (4)
Hepatocellular injury (Hepatobiliary disorders) | 2 (2) | 2 (3)

LIMITATIONS AND CAVEATS:
At the data cut-off date, treatment with rAd-IFN had not resulted in statistically significant differences from the control group (celecoxib + gemcitabine) in the primary efficacy endpoint (OS) or secondary efficacy endpoints. The study was powered to potentially show statistical significance with 300 patients enrolled. Only 82 patients were screened and 53 were randomised.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-12-11): https://cdn.clinicaltrials.gov/large-docs/76/NCT03710876/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-05): https://cdn.clinicaltrials.gov/large-docs/76/NCT03710876/SAP_001.pdf